CLINICAL TRIAL: NCT05033210
Title: Prevention of Mental Health Problems Among Persons Without Personal Housing in the Context of the COVID-19 Epidemic: a Randomized Controlled Trial
Brief Title: Prevention of Mental Health Problems Among Persons Without Personal Housing in the Context of the COVID-19 Epidemic
Acronym: RESPOND-FR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ANRS0065s
Record Dates: First submitted 2021-09-01; First posted 2021-09-02 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Psychological Distress; Quality of Life; Psychosocial Intervention
Keywords: Mental Health; Psychological Distress; COVID-19; Unstable Housing; Psychosocial interventions; Human Migration
MeSH Terms: conditions — Psychological Well-Being; COVID-19 | interventions — Psychological First Aid

STUDY DESIGN:
Intervention Model Description: After screening and baseline assessments, participants will be randomised to either the treatment group (n=105) or the comparison group (n=105), with an equal probability of assignment to each group (allocation ratio 1:1). The trial is a single-blind RCT (i.e. outcome assessors are blind to treatment allocation). Randomisation will be carried out through computerised software (Castor EDC) using limited block size (e.g. 6-12 participants per block) and will be performed by an independent person who is not involved in the assessment.
Who Masked: Outcomes Assessor
Masking Description: The statistical analysis will be masked, this means that the statistician will not know the treatment groups until the end of the analysis. In addition, this person will not be involved in the choice of the participants, the administration of the intervention, in study assessments or in data entry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The control group will receive Psychological First Aid (PFA) and Care as Usual (CAU)
  Interventions: Behavioral: Psychological First Aid (PFA); Behavioral: Care as Usual (CAU)
- Treatment Group (Experimental): The treatment group will receive the stepped-care program consisting of Doing What Matters (DWM) (step 1) and Problem Management Plus (PM+) (step 2), in addition to Psychological First Aid (PFA) and care as usual (CAU). Step 2 will only be provided if the participant still has elevated levels of psychological distress (K10 > 15.9) at 2 weeks after DWM, i.e. during the second quantitative assessment at 2 weeks after DWM.
  Interventions: Behavioral: Psychological First Aid (PFA); Behavioral: Care as Usual (CAU); Behavioral: Doing What Matters in Times of Stress (DWM); Behavioral: Problem Management Plus (PM+)

INTERVENTIONS:
Behavioral: Psychological First Aid (PFA) — PFA is a WHO developed support strategy that involves humane, supportive and practical help for individuals living in a serious humanitarian crisis. PFA does not necessarily involve a discussion of the event(s) that cause the distress but aims particularly at five basic elements that are crucial to promote in the aftermath of crises, i.e. a sense of safety, calm, self- and community efficacy, connectedness, and hope (Hobfoll et al., 2007). It consists of a conversation (approximately 30-45 minutes) that a helper has with a participant which can be provided remotely (e.g. videoconferencing or telephone). It has various themes; the helper provides non-intruding practical care and support, listen to needs and concerns, helps people to address basic needs (e.g. information), listens to people without pressuring them to talk, comforts people and helps them to feel calm, helps people to connect to information, services, and social support, and protects people from further harm (WHO, 2011).
Behavioral: Care as Usual (CAU) — In addition to PFA, both arms will be allowed to receive any usual care (CAU). CAU ranges from community care to specialised psychological treatments.
Behavioral: Doing What Matters in Times of Stress (DWM) — DWM is based on the acceptance and commitment therapy (ACT), a form of cognitive-behavioural therapy, with distinct features (Hayes, Levin, Plumb-Vilardaga, Villatte & Pistorello, 2013). ACT is based on the concept that ongoing attempts to suppress unwanted thoughts and feelings can make these problems worse, so instead it emphasises on learning new ways to accommodate these thoughts and feelings without letting them dominate. ACT has been shown to be useful for a range of mental health issues (Tjak et al., 2015) and has been used successfully in a guided self-help format (Hayes et al., 2013). DWM includes five sections (or modules), each of which focuses on a specific skill. In this study, the DWM program will be delivered as an online intervention. The DWM intervention, i.e. both the audios and the self-help guide, will be adapted for use on a smartphone or other device with internet access.
  Arms: Treatment Group
Behavioral: Problem Management Plus (PM+) — PM+ is a brief, psychological intervention program based on cognitive behavioural therapy (CBT) techniques that are empirically supported and formally recommended by the WHO (Dua et al., 2011). The manual involves the following empirically supported elements: problem solving plus stress management, behavioural activation, facing fears, and accessing social support. In these 90-minute sessions participants may talk to trained non-professional helpers (who are supervised by registered (clinical) psychologists). PM+ has four core features: it is brief (five sessions); delivered by non-specialist helpers; transdiagnostic thereby addressing depression, anxiety, PTSD, stress and problems as defined by people themselves; and originally designed for people in low-income country communities but easily adaptable to different (vulnerable) populations, cultures and languages.
  Arms: Treatment Group

SUMMARY:
The Covid-19 pandemic is having a great impact on the long-term mental health and well-being. Reports on the levels of psychological distress are concerning. This can be due to the pandemic, as well as social distancing, employment and economic consequences.

Healthcare workers, the elderly, youths, and persons experiencing socio-economic adversity are at risk of developing psychological distress. In this context, healthcare systems risk being overcharged, facing a growing demand.

Cognitive Behaviour Therapies managing psychological distress have been formally recommended. WHO has implemented different escalated psychosocial interventions, such as Problem Management Plus, PM+; Doing What Matters in Times of Stress, DWM; and Psychological First Aid, PFA. Their aim is to help individuals manage their stress in order to decrease the occurrence of psychological problems. They do not replace care for severe mental health disorders, but can prevent the deterioration of individuals' mental health.

PM+ has previously been found to be effective in situations of endemic conflict or violence in Pakistan and Kenya. The implementation of this program in Europe is being evaluated in the EU H2020 project STRENGHTS, focused in migrants from Syria. In the present trail, the investigators aim to further test its effectiveness in the context of psychological distress resulting from the COVID-19 pandemic.

Prior to the present trial, the investigators conducted a qualitative research study among potential beneficiaries and healthcare workers to evaluate the feasibility of DWM and PM+, which showed interest in stepped-care interventions in mental health, particularly if they are technology-based (mobile phones).

Our study is embedded in the larger, EU H2020 CORONAVIRUS-funded RESPOND project (Grant Agreement No 101016127). This project granted funding for a multicentric, single-blinded, randomised, controlled trial to evaluate the effectiveness of the stepped-care DWM and PM+ program vs. Care as Usual (CAU). In France, the investigators will focus on persons experiencing socioeconomic adversity, as defined by unstable housing conditions. A recent study showed that most of them are migrants. All subjects (210) will receive PFA and CAU. In addition to PFA and CAU, the treatment group (105 subjects) will receive the intervention DWM (with or without PM+). The primary outcome will be the decrease in symptoms of anxiety and depression from baseline to two-months follow-up.

DETAILED DESCRIPTION:
STUDY POPULATION Our population is composed of adults (18 years or older), with unstable housing status , speaking one of the languages of the research (Arabic, Dari, French or Pashto).

CALCULATION OF THE SAMPLE SIZE Based on prior studies (Bryant et al., 2017; Rahman et al., 2016b), the investigators aim to detect a small to medium Cohen's d effect size of 0.3 in the PM+ group at 2 months post-treatment based on the primary composite outcome PHQ-ADS (Kroenke et al., 2016; 2019). The PHQ-ADS is the combined sum score of depression and anxiety symptoms of the PHQ-9 and GAD-7, respectively and has shown good internal consistency (α = .88 to .92) (Kroenke et al., 2016; 2019). A power calculation for a repeated measurement design (with STATA) suggests a minimum sample size of N=73 per group (power=0.80, alpha=0.05, two-sided, rho=0.9). Considering 30% attrition, the investigators aim to include a total number of 210 participants (105 in the stepped-care DWM/PM+ treatment group (with PFA and CAU) and 105 in the PFA and CAU comparison group).

STATISTICAL METHODS The statistical analysis will estimate the effectiveness of the stepped-care programs DWM/PM+ intervention compared to PSP and CAU alone.

The primary outcome (PHQ-ADS scale) will be summarized using the number of subjects (n), minimum and maximum; and means, standard deviations (SD) for normally distributed data, or medians and interquartile ranges for non-normally distributed data. To measure comparisons at baseline between the two treatment groups t-tests (continuous variables) or chi-squared tests (categorical variables) will be conducted for normally distributed data; Mann-Whitney tests will be conducted for continuous non-normally distributed data. Health economic analysis will be conducted to determine the difference in costs and outcomes in the intervention arm as compared to the care as usual group. Primary analysis will be the total costs over the 2-month follow-up treatment period. Between-group comparison of mean costs will be completed using standard t-test with ordinary least squares regression used for adjusted analysis, with the validity of results confirmed using bootstrapping.

ETHICAL CONSIDERATIONS This study will fully comply with relevant European and national regulations concerning data protection, privacy regulations, and the procedures for obtaining informed consent.

* Informed consent Before being enrolled in the study, participants will be informed by the project manager and/or the main investigator about the aims and scope of the study in a form understandable to them. The individual will have one week to decide if it participates. If so, he/she will sign the consent form with the main investigator.
* Withdrawal of individual subjects Participants can leave the study at any time for any reason if they wish to do so without any consequences for them. The investigator can decide to withdraw a participant from the study for urgent medical reasons.

If a subject decides to withdraw from the study, the investigator will ask for the reason. Withdrawal from the study will have no effect on the regular treatment. Subjects who leave the study for medical reasons will be followed until the interfering condition has resolved or reached a stable state.

* Monitoring Monitoring includes review of helpers' records of PM+, supervision records including intervention fidelity monitoring and supervision of supervisors by the master trainers. The supervision of helpers will be scheduled weekly. The supervision will be given by the study psychologist. The supervising psychologist will also receive supervision from the master trainers and these supervisions will be scheduled monthly. Audio recordings on the form helpers make the interventions and pass the questionnaires will be taken. These records will assess as well the adherence to the interventions. Monitoring of the assessments will be the responsibility of the supervisor. In case of any concerns about the capacity of the assessors to carry out their roles, the project manager will conduct full assessments to ensure quality. This oversight will help ensure that any potential concerns about the capacity of assessors to carry out their roles is picked up and responded to.
* Benefits and risks of the research Participants randomized into the DWM/PM+ treatment group may benefit from their participation in terms of expected reductions in psychological distress. The risks associated with participation are estimated to be minimal, since DWM and PM+ reduced psychological distress in previous studies (Purgato et al., 2019; Tol et al., 2020; Bryant et al., 2017; Rahman et al., 2016b). Participants in both the treatment and comparison group will not be withheld care as usual.

It is possible that participants experience stress during the PM+ sessions. The intervention will be supervised and strictly monitored by experienced psychologists. If a participant deteriorates during the intervention period, (s)he can be referred to an external specialist (licensed psychologist or psychiatrist). Whenever referral has taken place, it will be actively followed-up by the researchers. In case of an undesirable emotional reaction either during the intervention or during follow-up assessments, the researchers and clinicians will be available to provide support if necessary.

If a participant has elevated symptoms of psychological distress in follow-up assessments, (s)he will be advised to contact his/her general practitioner (part of the CAU), who may refer the participant for continued or high-intensity treatment.

- Adverse events (AE) Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the trial procedure or to the stepped care DWM and PM+ intervention. All AEs reported spontaneously by the subject or observed by the investigator or his staff will be recorded. All AEs will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist.

• Compensation for injury

Participation in the study only carries negligible risks for the research subjects; therefore. An insurance has been taken by the study promotor to guarantee its civil responsibility, according to the French Public Health Code.

* Incentives Participants will also receive 60 euros (in vouchers) in total (20 euros on visit 1, 20 euros on visit 3, and 20 euros on visit 4).
* Data management All data will be handled confidentially and will be coded by a code known only to the research team. Processing of personal data will comply with the General Data Regulation (GDPR). Additionally, this study adheres to the Research Data Management Policy of the ANRS.

Data including personal information will be stored in a locked file at INSERM to ensure the confidentiality of the study participants. Only authorized research personnel will have access to these data. According to the data management rules of RESPOND, all partners acknowledge and agree that no personal data, as defined in Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC (GDPR), will be exchanged between the Parties. Moreover, all partners in RESPOND acknowledge and agree that each partner is considered an independent controller, as defined in GDPR, for its processing of personal data and will act in accordance with applicable data protection laws (including but not limited to GDPR).

ELIGIBILITY:
Inclusion Criteria:

Participants will have to be 18 years or older, without stable housing, meet the criteria for psychological distress (K10 > 15.9), speak one of the study languages (Arabic, French, Pashto, Dari) and agree to participate in the study.

Exclusion Criteria:

Individuals with an acute medical or psychiatric condition requiring urgent medical services, at risk for suicide, with moderate/severe cognitive impairment (e.g., severe intellectual disability or dementia), under juridical protection (guardianship, tutorship, legal safeguard), with a psychotropic treatment whose dose has changed during the last 2 months, or refusing to participate in the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
PHQ-ADS | Week 2, Week 8, Week 14, Week 22
  The PHQ-ADS is the sum of the PHQ-9 and GAD-7 scores (details of both instruments summarised below) and thus can range from 0 to 48, with higher scores indicating higher levels of depression and anxiety symptomatology. Two validation studies of the PHQ-ADS in trial data-sets of patients with chronic (musculoskeletal) pain and oncological diseases have been published (Kroenke et al., 2016; Kroenke et al., 2019). Evidence shows high internal reliability (Cronbach's alpha of 0.8 to 0.9), strong convergent and construct validity, sufficient uni-dimensionality and evidence for sensitivity to change (i.e. differentiating between individuals classified as worse, stable, or improved by a reference measure at three months post-intervention).

SECONDARY OUTCOMES:
Level of depression (PHQ-9) | Week 2, Week 8, Week 14, Week 22
  Depressive symptoms during the past two weeks will be measured using the Patient Health Questionnaire depressive module. It asks how often someone was bothered by each of the nine DSM-5 criteria and scores answers on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day) (Kroenke, Spitzer, & Williams, 2001). In addition to the nine items, the PHQ-9 asks: "If you checked off any problems, how difficult have these problems made it for you to do your work, take care of things at home, or get along with other people?", which is to be answered with "Not difficult at all", "Somewhat difficult", "Very difficult", or "Extremely difficult". For the current study, changes in caseness in depression will be examined. A cut-off score of 10 will be used, which has been found to be a valid cut-off point for diagnosis (Manea, Gilbody & McMillan, 2021).
Level of anxiety (GAD-7) | Week 2, Week 8, Week 14, Week 22
  The Generalized Anxiety Disorder (GAD-7) questionnaire is a seven-item, self-report anxiety questionnaire which assesses the degree to which the patient has been bothered by feeling nervous, anxious or on edge over the last two weeks. Items also include other generalised anxiety symptoms such as being unable to stop worrying about multiple things, having trouble relaxing or sitting still, feeling irritable and being afraid of something bad happening at all times (Spitzer et al., 2006). Items are scored from 0 to 3, respectively for experiencing symptoms 'not at all', for 'several days', for 'more than half the days' and for 'nearly every day'. The total score ranges from 0 to 21. Cut-off points for mild, moderate and severe anxiety are scores of 5, 10 and 15, respectively (Spitzer et al., 2006). A score of 10 has been identified as the optimal cut-off score to balance specificity and sensitivity (Spitzer et al., 2006).
Severity of posttraumatic stress disorder (PCL-5) | Week 2, Week 8, Week 14, Week 22
  Posttraumatic stress disorder (PTSD) symptoms during the past week according to the DSM-5 PTSD diagnosis will be measured using the PTSD Checklist for DSM-5 (PCL-5) (Weathers et al., 2013). A shortened 8-item version of the original PCL-5 (a 20-item checklist which corresponds with the 20 DSM-5 PTSD symptoms) will be used. Items are rated on a 0-4 scale. Added up, the maximum severity score is 32. Higher scores indicate higher symptomatology. In a comparison of two abbreviated versions, i.e., the 4-item and 8-item versions of the PCL-5, the PCL-5 8 item version showed a strong correlation with the total scale, greater internal consistency, and allowed for sufficient variability in patient response. There were no significant differences in the sensitivity and specificity between the total 20-item PCL-5 scale and the 8-item scale (Price et al., 2016).
Self-identified problems (PSYCHLOPS) | Week 2, Week 8, Week 14, Week 22
  The Psychological Outcomes Profiles (PSYCHLOPS) scale is a patient-generated outcome measure as an indicator of change after therapy (Ashworth et al., 2004). PSYCHLOPS consists of four questions. It contains three domains: problems (2 questions), function (1 question), and wellbeing (1 question). Participants are asked to give free text responses to the problem and function domains. Responses are scored on an ordinal six-point scale producing a maximum score of 18 (six points per domain). PSYCHLOPS has been validated in primary care populations across several countries (Czachowski, Seed, Schofield, & Ashworth, 2011; Héðinsson, Kristjánsdóttir, Ólason, & Sigurðsson, 2013).
Psychotic symptoms (MINI) | Week 2, Week 8, Week 14, Week 22
  M.I.N.I is a structured diagnostic interview, validated in French (Sheehan et al., 1998), which explores in a standardised manner the main psychiatric troubles which appear in the first axis of the DSM-IV (American Psychiatric Association, 1994). We will use questions 1 to 7 from Item L (psychotic troubles), to determine the presence of psychotic symptoms during the last 6 months.
Resilience based on exposure to stressful events, general and COVID-19 related (MIMIS) | Week 2, Week 8, Week 14, Week 22
  The Mainz Inventory of Microstressors (MIMIS) was recently developed to measure objective microstressors of modern life in the past 7 days (Chmitorz et al., 2020). In the Dynacore-C study (Veer et al., 2021) this was changed into a period of 2 weeks and a shorter general and COVID-19 specific stressor list. The MIMIS uses a definition of resilience as a trade-off between the outcome of mental health and exposure to adversity. Outcome-based resilience will be assessed by relating self-reported changes in mental health problems (i.e. anxiety and depression) over the past 2 weeks (assessed with the PHQ-ADS) to the self-reported exposure to 11 categories of general stressors (life events and daily stressors such as physical health problems, family conflicts or separation form a loved one) and 29 COVID-19 crisis related stressors (such as COVID-19 symptoms, belonging to a risk group for serious COVID-19 symptoms, loss of social contact, or problems arranging childcare (Veer et al., 2021).
Quality of life (EQ-5D-5L) | Week 2, Week 8, Week 14, Week 22
  The EQ-5D-5L measures quality of life and consists of two parts, the EQ-5D and the EQ VAS. Part 1, the EQ-5D, rates the level of impairment across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ-5D-5L is an adapted version of the EQ-5D(-3L), which only had three response options for each dimensions and was therefore thought to not sufficiently capture milder health issues and small changes between different states of health (Herdman et al., 2011).
Cost of care: impact on use of health system, other services, time out of employment and other usual activities and need for informal care (CSRI) | Week 2, Week 8, Week 14, Week 22
  The Client Service Receipt Inventory (CSRI) was developed for the collection of data on service utilization (e.g. use of health system, other services, time out of employment and other usual activities, need for informal care) and related characteristics of people with mental disorders, as the basis for calculating the costs of care for mental health cost-effectiveness research.
Resilience factors: a positive approach (PASSc) | Week 2, Week 14, Week 22
  PASSc is based on a positive approach to resilience theory (PASTOR; Kalisch et al, 2015; Kalisch et al, 2021). PASTOR theory conceptualizes resilience as an outcome: the maintenance of mental health after exposure to a stressor. The positive approach would no longer be measured as resilience, but as a resilience factor. She wants to capture the mechanism leading to this resilience.

OTHER OUTCOMES:
Socio-demographic information | Week 2, Week 8, Week 14, Week 22
  Socio-demographic information will be collected with predefined items based on the REDEFINE and STRENGTHS studies (i.e. age, gender, nationality, years of education, relationship status, and main work-status and additional questions regarding country of birth, household population (incl. children < 18 and elderly people), household income on average, occupational area working, mental health condition and overall current health status and housing (square meters of the house, outdoor space available).
BTQ: Brief Trauma Questionnaire | Week 2, Week 14, Week 22
  Brief self-report questionnaire derived from the Brief Trauma Interview (Schnurr et al., 1995). BTQ is designed to assess traumatic exposure. It provides a comprehensive assessment of DSM V Criterion A (stressors), of which exposure to trauma is an example.
Treatment fidelity | Weeks 3 to 7, 9 to 13
  Process monitoring of the full stepped-care intervention includes review of helpers' records of DWM phone calls and PM+ sessions with clients; helpers' supervision records including intervention fidelity monitoring, and supervision of supervisors by intervention trainers. To monitor treatment fidelity of DWM, participants' usage of the DWM app will be tracked. To monitor treatment fidelity of PM+, treatment sessions will be audio-recorded. If participants are randomized into the treatment group, they will be asked for a separate consent to record the sessions. Giving consent to the audio recording is no requirement to receive the PM+ program.
Satisfaction and acceptability DWM/PM+ | Week 8, Week 14
  Satisfaction and acceptability of the stepped-care DWM/PM+ intervention is measured through qualitative process evaluation. Additionally, at the first assessment after DWM (T2) and after PM+ (T3), participants will also fill out a questionnaire to measure their satisfaction with the intervention. The CSQ-I for the web-based intervention DWM (Boss et al., 2016) and the CSQ-8 for PM+ Client Satisfaction Questionnaire (CSQ-8; Attkisson & Zwick, 1982)
Events related to the COVID-19 pandemic | Week 2, Week 8, Week 14, Week 22
  We ask participants about events they have experienced in connection with the COVID-19 pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tortelli, Doctor, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Maria Melchior, Doctor, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- France (2):
  - Normandy Psychotrauma Center, Caen, Normandy
  - CAPSYS, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie results in a publication will be shared on the RESPOND website (https://respond-project.eu/). At the end of the randomised trial, other meta-analysis can be conducted in the framework of research with individuals in unstable housing. For this reason, all data will be stocked during 15 years by the sponsor of the research (ANRS|MIE) and the investigator centre (INSERM).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from the end of the research and will be stored during 15 years.
Access Criteria: Data will be shared with the different partners of the RESPOND Project through CASTOR EDC to conduct different analysis even after the end of the research project. Each individual having access to CASTOR will have its own password, and the rights of every user of this software in a particular country will be decided by the project manager of that country.

REFERENCES:
- [Background] A-Tjak JG, Davis ML, Morina N, Powers MB, Smits JA, Emmelkamp PM. A meta-analysis of the efficacy of acceptance and commitment therapy for clinically relevant mental and physical health problems. Psychother Psychosom. 2015;84(1):30-6. doi: 10.1159/000365764. Epub 2014 Dec 24. PMID 25547522
- [Background] Altman DG. Endorsement of the CONSORT statement by high impact medical journals: survey of instructions for authors. BMJ. 2005 May 7;330(7499):1056-7. doi: 10.1136/bmj.330.7499.1056. No abstract available. PMID 15879389
- [Background] Ashbaugh AR, Houle-Johnson S, Herbert C, El-Hage W, Brunet A. Psychometric Validation of the English and French Versions of the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). PLoS One. 2016 Oct 10;11(10):e0161645. doi: 10.1371/journal.pone.0161645. eCollection 2016. PMID 27723815
- [Background] Ashworth M, Shepherd M, Christey J, Matthews V, Wright K, Parmentier H, et al. A client-generated psychometric instrument: The development of 'PSYCHLOPS.' Couns Psychother Res [Internet]. 2004;4(2):27-31. Available from: https://www.tandfonline.com/doi/abs/10.1080/14733140412331383913
- [Background] Baggaley RF, Ganaba R, Filippi V, Kere M, Marshall T, Sombie I, Storeng KT, Patel V. Detecting depression after pregnancy: the validity of the K10 and K6 in Burkina Faso. Trop Med Int Health. 2007 Oct;12(10):1225-9. doi: 10.1111/j.1365-3156.2007.01906.x. PMID 17956505
- [Background] Baillie AJ. Predictive gender and education bias in Kessler's psychological distress Scale (k10). Soc Psychiatry Psychiatr Epidemiol. 2005 Sep;40(9):743-8. doi: 10.1007/s00127-005-0935-9. Epub 2005 Sep 5. PMID 16142511
- [Background] Banbury A, Nancarrow S, Dart J, Gray L, Parkinson L. Telehealth Interventions Delivering Home-based Support Group Videoconferencing: Systematic Review. J Med Internet Res. 2018 Feb 2;20(2):e25. doi: 10.2196/jmir.8090. PMID 29396387
- [Background] Blavatnik School of Government University of Oxford,
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Boyd L, Baker E, Reilly J. Impact of a progressive stepped care approach in an improving access to psychological therapies service: An observational study. PLoS One. 2019 Apr 9;14(4):e0214715. doi: 10.1371/journal.pone.0214715. eCollection 2019. PMID 30964883
- [Background] Bryant RA, Schafer A, Dawson KS, Anjuri D, Mulili C, Ndogoni L, Koyiet P, Sijbrandij M, Ulate J, Harper Shehadeh M, Hadzi-Pavlovic D, van Ommeren M. Effectiveness of a brief behavioural intervention on psychological distress among women with a history of gender-based violence in urban Kenya: A randomised clinical trial. PLoS Med. 2017 Aug 15;14(8):e1002371. doi: 10.1371/journal.pmed.1002371. eCollection 2017 Aug. PMID 28809935
- [Background] Busch-Geertsema V, Edgar W. Homelessness and homeless policies in Europe: Lessons from research [Internet]. Brussels; 2010. Available from: http://www.sociallabel.be/sites/default/files/doc/116829_pod_broch_homelessnes_eng_v3_0.pdf
- [Background] Cambridge University Press. Bootstrap Methods and Their Applications. Cambridge; 1997. 582 p.
- [Background] Campion J, Bhugra D, Bailey S, Marmot M. Inequality and mental disorders: opportunities for action. Lancet. 2013 Jul 20;382(9888):183-4. doi: 10.1016/S0140-6736(13)61411-7. No abstract available. PMID 23870520
- [Background] Chisholm D, Knapp MR, Knudsen HC, Amaddeo F, Gaite L, van Wijngaarden B. Client Socio-Demographic and Service Receipt Inventory--European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: Inputs Linked to Outcome Domains and Needs. Br J Psychiatry Suppl. 2000;(39):s28-33. doi: 10.1192/bjp.177.39.s28. PMID 10945075
- [Background] Chmitorz A, Kurth K, Mey LK, Wenzel M, Lieb K, Tuscher O, Kubiak T, Kalisch R. Assessment of Microstressors in Adults: Questionnaire Development and Ecological Validation of the Mainz Inventory of Microstressors. JMIR Ment Health. 2020 Feb 24;7(2):e14566. doi: 10.2196/14566. PMID 32130154
- [Background] Cohen S, Williamson G. Perceived stress in a probability sample of the United States [Internet]. Vol. 13, The Social Psychology of Health. 1988. p. 31-67. Available from: http://doi.apa.org/psycinfo/1988-98838-002
- [Background] Cuijpers P, Munoz RF, Clarke GN, Lewinsohn PM. Psychoeducational treatment and prevention of depression: the "Coping with Depression" course thirty years later. Clin Psychol Rev. 2009 Jul;29(5):449-58. doi: 10.1016/j.cpr.2009.04.005. Epub 2009 Apr 18. PMID 19450912
- [Background] Czachowski S, Seed P, Schofield P, Ashworth M. Measuring psychological change during cognitive behaviour therapy in primary care: a Polish study using 'PSYCHLOPS' (Psychological Outcome Profiles). PLoS One. 2011;6(12):e27378. doi: 10.1371/journal.pone.0027378. Epub 2011 Dec 15. PMID 22194783
- [Background] Dawson KS, Schafer A, Anjuri D, Ndogoni L, Musyoki C, Sijbrandij M, van Ommeren M, Bryant RA. Feasibility trial of a scalable psychological intervention for women affected by urban adversity and gender-based violence in Nairobi. BMC Psychiatry. 2016 Nov 18;16(1):410. doi: 10.1186/s12888-016-1117-x. PMID 27863515
- [Background] de Graaff AM, Cuijpers P, Acarturk C, Bryant R, Burchert S, Fuhr DC, Huizink AC, de Jong J, Kieft B, Knaevelsrud C, McDaid D, Morina N, Park AL, Uppendahl J, Ventevogel P, Whitney C, Wiedemann N, Woodward A, Sijbrandij M. Effectiveness of a peer-refugee delivered psychological intervention to reduce psychological distress among adult Syrian refugees in the Netherlands: study protocol. Eur J Psychotraumatol. 2020 Jan 20;11(1):1694347. doi: 10.1080/20008198.2019.1694347. eCollection 2020. PMID 32082506
- [Background] Department of Mental Health and Substance Abuse. PROBLEM MANAGEMENT PLUS (PM+): Individual psychological help for adults impaired by distress in communities exposed to adversity [Internet]. Geneva; 2016. Available from: https://www.who.int/publications/i/item/WHO-MSD-MER-16.2%0Awww.who.int
- [Background] den Boer PC, Wiersma D, Van den Bosch RJ. Why is self-help neglected in the treatment of emotional disorders? A meta-analysis. Psychol Med. 2004 Aug;34(6):959-71. doi: 10.1017/s003329170300179x. PMID 15554567
- [Background] Department of Mental Health and Substance Abuse. Scalable psychological interventions for people in communities affected by adversity. A new area of mental health and psychosocial work at WHO [Internet]. 2017. Available from: https://apps.who.int/iris/handle/10665/254581
- [Background] Donker T, Comijs H, Cuijpers P, Terluin B, Nolen W, Zitman F, Penninx B. The validity of the Dutch K10 and extended K10 screening scales for depressive and anxiety disorders. Psychiatry Res. 2010 Mar 30;176(1):45-50. doi: 10.1016/j.psychres.2009.01.012. Epub 2010 Jan 13. PMID 20071036
- [Background] Donker T, van Straten A, Marks I, Cuijpers P. Quick and easy self-rating of Generalized Anxiety Disorder: validity of the Dutch web-based GAD-7, GAD-2 and GAD-SI. Psychiatry Res. 2011 Jun 30;188(1):58-64. doi: 10.1016/j.psychres.2011.01.016. Epub 2011 Feb 19. PMID 21339006
- [Background] Dragan M, Grajewski P, Shevlin M. Adjustment disorder, traumatic stress, depression and anxiety in Poland during an early phase of the COVID-19 pandemic. Eur J Psychotraumatol. 2021 Jan 26;12(1):1860356. doi: 10.1080/20008198.2020.1860356. eCollection 2021. PMID 34992743
- [Background] Dua T, Barbui C, Clark N, Fleischmann A, Poznyak V, van Ommeren M, Yasamy MT, Ayuso-Mateos JL, Birbeck GL, Drummond C, Freeman M, Giannakopoulos P, Levav I, Obot IS, Omigbodun O, Patel V, Phillips M, Prince M, Rahimi-Movaghar A, Rahman A, Sander JW, Saunders JB, Servili C, Rangaswamy T, Unutzer J, Ventevogel P, Vijayakumar L, Thornicroft G, Saxena S. Evidence-based guidelines for mental, neurological, and substance use disorders in low- and middle-income countries: summary of WHO recommendations. PLoS Med. 2011 Nov;8(11):e1001122. doi: 10.1371/journal.pmed.1001122. Epub 2011 Nov 15. PMID 22110406
- [Background] Edgar, B., Doherty, J. & Meert, H. 2004. Immigration And Homelessness In Europe, Policy Press.
- [Background] Epping-Jordan JE, Harris R, Brown FL, Carswell K, Foley C, Garcia-Moreno C, Kogan C, van Ommeren M. Self-Help Plus (SH+): a new WHO stress management package. World Psychiatry. 2016 Oct;15(3):295-296. doi: 10.1002/wps.20355. No abstract available. PMID 27717271
- [Background] Fledderus M, Bohlmeijer ET, Pieterse ME, Schreurs KM. Acceptance and commitment therapy as guided self-help for psychological distress and positive mental health: a randomized controlled trial. Psychol Med. 2012 Mar;42(3):485-95. doi: 10.1017/S0033291711001206. Epub 2011 Jul 11. PMID 21740624
- [Background] Foa, E. B. (1995) Posttraumatic stress diagnostic scale (PDS);, Minneapolis: National Computer Systems.
- [Background] Galenkamp H, Stronks K, Snijder MB, Derks EM. Measurement invariance testing of the PHQ-9 in a multi-ethnic population in Europe: the HELIUS study. BMC Psychiatry. 2017 Oct 24;17(1):349. doi: 10.1186/s12888-017-1506-9. PMID 29065874
- [Background] Gambin M, Sekowski M, Wozniak-Prus M, Wnuk A, Oleksy T, Cudo A, Hansen K, Huflejt-Lukasik M, Kubicka K, Lys AE, Gorgol J, Holas P, Kmita G, Lojek E, Maison D. Generalized anxiety and depressive symptoms in various age groups during the COVID-19 lockdown in Poland. Specific predictors and differences in symptoms severity. Compr Psychiatry. 2021 Feb;105:152222. doi: 10.1016/j.comppsych.2020.152222. Epub 2020 Dec 25. PMID 33388494
- [Background] Gandubert C, Scali J, Ancelin ML, Carriere I, Dupuy AM, Bagnolini G, Ritchie K, Sebanne M, Martrille L, Baccino E, Hermes A, Attal J, Chaudieu I. Biological and psychological predictors of posttraumatic stress disorder onset and chronicity. A one-year prospective study. Neurobiol Stress. 2016 Feb 4;3:61-67. doi: 10.1016/j.ynstr.2016.02.002. eCollection 2016 Jun. PMID 27981178
- [Background] Garcy AM, Vagero D. Unemployment and suicide during and after a deep recession: a longitudinal study of 3.4 million Swedish men and women. Am J Public Health. 2013 Jun;103(6):1031-8. doi: 10.2105/AJPH.2013.301210. Epub 2013 Apr 18. PMID 23597379
- [Background] Gurría A. Virtual 2020 G20 Digital Ministers Summit on COVID-19. Vol. April. Paris: OECD; 2020.
- [Background] Hayes SC, Levin ME, Plumb-Vilardaga J, Villatte JL, Pistorello J. Acceptance and commitment therapy and contextual behavioral science: examining the progress of a distinctive model of behavioral and cognitive therapy. Behav Ther. 2013 Jun;44(2):180-98. doi: 10.1016/j.beth.2009.08.002. Epub 2011 Jun 1. PMID 23611068
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Hinz A, Klein AM, Brahler E, Glaesmer H, Luck T, Riedel-Heller SG, Wirkner K, Hilbert A. Psychometric evaluation of the Generalized Anxiety Disorder Screener GAD-7, based on a large German general population sample. J Affect Disord. 2017 Mar 1;210:338-344. doi: 10.1016/j.jad.2016.12.012. Epub 2016 Dec 18. PMID 28088111
- [Background] Ho FY, Yeung WF, Ng TH, Chan CS. The Efficacy and Cost-Effectiveness of Stepped Care Prevention and Treatment for Depressive and/or Anxiety Disorders: A Systematic Review and Meta-Analysis. Sci Rep. 2016 Jul 5;6:29281. doi: 10.1038/srep29281. PMID 27377429
- [Background] Hobfoll SE, Watson P, Bell CC, Bryant RA, Brymer MJ, Friedman MJ, Friedman M, Gersons BP, de Jong JT, Layne CM, Maguen S, Neria Y, Norwood AE, Pynoos RS, Reissman D, Ruzek JI, Shalev AY, Solomon Z, Steinberg AM, Ursano RJ. Five essential elements of immediate and mid-term mass trauma intervention: empirical evidence. Psychiatry. 2007 Winter;70(4):283-315; discussion 316-69. doi: 10.1521/psyc.2007.70.4.283. PMID 18181708
- [Background] Marshall C. The inter-agency standing committee (IASC) guidelines on mental health and psychosocial support (MHPSS) in emergency settings: a critique. Int Rev Psychiatry. 2022 Sep;34(6):604-612. doi: 10.1080/09540261.2022.2147420. Epub 2022 Dec 11. PMID 36502397
- [Background] Kertz S, Bigda-Peyton J, Bjorgvinsson T. Validity of the Generalized Anxiety Disorder-7 scale in an acute psychiatric sample. Clin Psychol Psychother. 2013 Sep-Oct;20(5):456-64. doi: 10.1002/cpp.1802. Epub 2012 May 17. PMID 22593009
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Kroenke K, Baye F, Lourens SG. Comparative validity and responsiveness of PHQ-ADS and other composite anxiety-depression measures. J Affect Disord. 2019 Mar 1;246:437-443. doi: 10.1016/j.jad.2018.12.098. Epub 2018 Dec 25. PMID 30599366
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Wu J, Yu Z, Bair MJ, Kean J, Stump T, Monahan PO. Patient Health Questionnaire Anxiety and Depression Scale: Initial Validation in Three Clinical Trials. Psychosom Med. 2016 Jul-Aug;78(6):716-27. doi: 10.1097/PSY.0000000000000322. PMID 27187854
- [Background] Lace JW, Greif TR, McGrath A, Grant AF, Merz ZC, Teague CL, et al. Investigating the factor structure of the K10 and identifying cutoff scores denoting nonspecific psychological distress and need for treatment. Ment Heal Prev [Internet]. 2019;13(January):100-6. Available from: https://doi.org/10.1016/j.mhp.2019.01.008
- [Background] Lamers F, Jonkers CC, Bosma H, Penninx BW, Knottnerus JA, van Eijk JT. Summed score of the Patient Health Questionnaire-9 was a reliable and valid method for depression screening in chronically ill elderly patients. J Clin Epidemiol. 2008 Jul;61(7):679-87. doi: 10.1016/j.jclinepi.2007.07.018. Epub 2008 Feb 14. PMID 18538262
- [Background] Le Méner E, Oppenchaim N. The Temporary Accommodation of Homeless Families in Ile-de-France: Between Social Emergency and Immigration Management 1. Eur J Homelessness [Internet]. 2012;6(1):83-103. Available from: https://www.feantsaresearch.org/download/article-4-31158086039476347447.pdf
- [Background] Legleye S, Karila L, Beck F, Reynaud M. Validation of the CAST, a general population Cannabis Abuse Screening Test. J Subst Use [Internet]. 2007;12(4):233-42. Available from: https://www.tandfonline.com/doi/abs/10.1080/14659890701476532
- [Background] Longchamps C, Ducarroz S, Crouzet L, El Aarbaoui T, Allaire C, Colleville A-C, et al. Connaissances, attitudes et pratiques liées à L'épidémie de Covid-19 et son impact chez les personnes en situation de précarité vivant en centre d'hébergement en France : Premiers Résultats de l'étude Echo. BEH [Internet]. 2021;(1):2-9. Available from: http://beh.santepubliquefrance.fr/beh/2021/Cov_1/2021_Cov_1_1.html
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Manea L, Gilbody S, McMillan D. Optimal cut-off score for diagnosing depression with the Patient Health Questionnaire (PHQ-9): a meta-analysis. CMAJ. 2012 Feb 21;184(3):E191-6. doi: 10.1503/cmaj.110829. Epub 2011 Dec 19. PMID 22184363
- [Background] McGinty EE, Presskreischer R, Han H, Barry CL. Psychological Distress and Loneliness Reported by US Adults in 2018 and April 2020. JAMA. 2020 Jul 7;324(1):93-94. doi: 10.1001/jama.2020.9740. PMID 32492088
- [Background] Morgan C, Knowles G, Hutchinson G. Migration, ethnicity and psychoses: evidence, models and future directions. World Psychiatry. 2019 Oct;18(3):247-258. doi: 10.1002/wps.20655. PMID 31496097
- [Background] Murray LK, Dorsey S, Bolton P, Jordans MJ, Rahman A, Bass J, Verdeli H. Building capacity in mental health interventions in low resource countries: an apprenticeship model for training local providers. Int J Ment Health Syst. 2011 Nov 18;5(1):30. doi: 10.1186/1752-4458-5-30. PMID 22099582
- [Background] Nose M, Ballette F, Bighelli I, Turrini G, Purgato M, Tol W, Priebe S, Barbui C. Psychosocial interventions for post-traumatic stress disorder in refugees and asylum seekers resettled in high-income countries: Systematic review and meta-analysis. PLoS One. 2017 Feb 2;12(2):e0171030. doi: 10.1371/journal.pone.0171030. eCollection 2017. PMID 28151992
- [Background] Okruszek L, Aniszewska-Stanczuk A, Piejka A, Wisniewska M, Zurek K. Safe but Lonely? Loneliness, Anxiety, and Depression Symptoms and COVID-19. Front Psychol. 2020 Dec 4;11:579181. doi: 10.3389/fpsyg.2020.579181. eCollection 2020. PMID 33343454
- [Background] Organisation Mondiale de la Santé. Gestion des problèmes Plus (PM+). Soutien psychosocial individuel pour adultes affectés par la détresse dans les communautés exposées à l'adversité [Internet]. Geneva; 2018. Available from: https://apps.who.int/iris/handle/10665/275831
- [Background] Organisation Mondiale de la Santé. Faire ce qui compte en période de stress : Un guide illustré [Internet]. Geneva: World Health Organisation; 2020. 132 p. Available from: https://cdn.who.int/media/docs/default-source/mental-health/sh-2020-fre-5-web.pdf?sfvrsn=90a35ada_2
- [Background] Organisation Mondiale de la santé, War Trauma Foundation, World Vision International. Les premiers secours psychologiques guide pour les travailleurs humanitaires sur le terrain [Internet]. Geneva; 2012. Available from: https://apps.who.int/iris/handle/10665/44779
- [Background] Pomerleau CS, Majchrzak MJ, Pomerleau OF. Nicotine dependence and the Fagerstrom Tolerance Questionnaire: a brief review. J Subst Abuse. 1989;1(4):471-7. PMID 2485293
- [Background] Price M, Szafranski DD, van Stolk-Cooke K, Gros DF. Investigation of abbreviated 4 and 8 item versions of the PTSD Checklist 5. Psychiatry Res. 2016 May 30;239:124-30. doi: 10.1016/j.psychres.2016.03.014. Epub 2016 Mar 8. PMID 27137973
- [Background] Public Health England. Disparities in the risk and outcomes of COVID-19 [Internet]. PHE Publications. London; 2020. Available from: https://www.gov.uk/government/publications/covid-19-review-of-disparities-in-risks-and-outcomes
- [Background] Purgato M, Carswell K, Acarturk C, Au T, Akbai S, Anttila M, Baumgartner J, Bailey D, Biondi M, Bird M, Churchill R, Eskici S, Hansen LJ, Heron P, Ilkkursun Z, Kilian R, Koesters M, Lantta T, Nose M, Ostuzzi G, Papola D, Popa M, Sijbrandij M, Tarsitani L, Tedeschi F, Turrini G, Uygun E, Valimaki MA, Wancata J, White R, Zanini E, Cuijpers P, Barbui C, Van Ommeren M. Effectiveness and cost-effectiveness of Self-Help Plus (SH+) for preventing mental disorders in refugees and asylum seekers in Europe and Turkey: study protocols for two randomised controlled trials. BMJ Open. 2019 May 14;9(5):e030259. doi: 10.1136/bmjopen-2019-030259. PMID 31092670
- [Background] Puric D, Vukcevic Markovic M. Development and validation of the Stressful Experiences in Transit Questionnaire (SET-Q) and its Short Form (SET-SF). Eur J Psychotraumatol. 2019 May 16;10(1):1611091. doi: 10.1080/20008198.2019.1611091. eCollection 2019. PMID 31164967
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Background] Rahman A, Riaz N, Dawson KS, Usman Hamdani S, Chiumento A, Sijbrandij M, Minhas F, Bryant RA, Saeed K, van Ommeren M, Farooq S. Problem Management Plus (PM+): pilot trial of a WHO transdiagnostic psychological intervention in conflict-affected Pakistan. World Psychiatry. 2016 Jun;15(2):182-3. doi: 10.1002/wps.20312. No abstract available. PMID 27265713
- [Background] Rutter LA, Brown TA. Psychometric Properties of the Generalized Anxiety Disorder Scale-7 (GAD-7) in Outpatients with Anxiety and Mood Disorders. J Psychopathol Behav Assess. 2017 Mar;39(1):140-146. doi: 10.1007/s10862-016-9571-9. Epub 2016 Sep 10. No abstract available. PMID 28260835
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Seeman TE, Singer BH, Rowe JW, Horwitz RI, McEwen BS. Price of adaptation--allostatic load and its health consequences. MacArthur studies of successful aging. Arch Intern Med. 1997 Oct 27;157(19):2259-68. PMID 9343003
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Shim RS, Compton MT. The Social Determinants of Mental Health: Psychiatrists' Roles in Addressing Discrimination and Food Insecurity. Focus (Am Psychiatr Publ). 2020 Jan;18(1):25-30. doi: 10.1176/appi.focus.20190035. Epub 2020 Jan 24. PMID 32047394
- [Background] Shoeb M, Weinstein H, Mollica R. The Harvard trauma questionnaire: adapting a cross-cultural instrument for measuring torture, trauma and posttraumatic stress disorder in Iraqi refugees. Int J Soc Psychiatry. 2007 Sep;53(5):447-63. doi: 10.1177/0020764007078362. PMID 18018666
- [Background] Sijbrandij M, Horn R, Esliker R, O'May F, Reiffers R, Ruttenberg L, Stam K, de Jong J, Ager A. The Effect of Psychological First Aid Training on Knowledge and Understanding about Psychosocial Support Principles: A Cluster-Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Jan 11;17(2):484. doi: 10.3390/ijerph17020484. PMID 31940865
- [Background] Smits N, Smit F, Cuijpers P, De Graaf R. Using decision theory to derive optimal cut-off scores of screening instruments: an illustration explicating costs and benefits of mental health screening. Int J Methods Psychiatr Res. 2007;16(4):219-29. doi: 10.1002/mpr.230. PMID 18188835
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Staufenbiel SM, Penninx BW, de Rijke YB, van den Akker EL, van Rossum EF. Determinants of hair cortisol and hair cortisone concentrations in adults. Psychoneuroendocrinology. 2015 Oct;60:182-94. doi: 10.1016/j.psyneuen.2015.06.011. Epub 2015 Jun 25. PMID 26176863
- [Background] Sterling P, Eyer J. Biological basis of stress-related mortality. Soc Sci Med E. 1981 Feb;15(1):3-42. doi: 10.1016/0271-5384(81)90061-2. No abstract available. PMID 7020084
- [Background] Stickley A, Koyanagi A. Loneliness, common mental disorders and suicidal behavior: Findings from a general population survey. J Affect Disord. 2016 Jun;197:81-7. doi: 10.1016/j.jad.2016.02.054. Epub 2016 Mar 2. PMID 26971125
- [Background] Sulaiman-Hill CM, Thompson SC. Selecting instruments for assessing psychological wellbeing in Afghan and Kurdish refugee groups. BMC Res Notes. 2010 Sep 8;3:237. doi: 10.1186/1756-0500-3-237. PMID 20825681
- [Background] Suri H. Purposeful sampling in qualitative research synthesis. Qual Res J [Internet]. 2011;11(2):63-75. Available from: https://www.emerald.com/insight/content/doi/10.3316/QRJ1102063/full/html#loginreload
- [Background] Thabet AA, Abu Tawahina A, El Sarraj E, Vostanis P. Exposure to war trauma and PTSD among parents and children in the Gaza strip. Eur Child Adolesc Psychiatry. 2008 Jun;17(4):191-9. doi: 10.1007/s00787-007-0653-9. PMID 18365135
- [Background] Young H, Harvey P. The sphere project: the humanitarian charter and minimum standards in disaster response: introduction. Disasters. 2004 Jun;28(2):99. doi: 10.1111/j.0361-3666.2004.00245.x. No abstract available. PMID 20958782
- [Background] Thomson RM, Katikireddi SV. Mental health and the jilted generation: Using age-period-cohort analysis to assess differential trends in young people's mental health following the Great Recession and austerity in England. Soc Sci Med. 2018 Oct;214:133-143. doi: 10.1016/j.socscimed.2018.08.034. Epub 2018 Aug 29. PMID 30195100
- [Background] Tol WA, Leku MR, Lakin DP, Carswell K, Augustinavicius J, Adaku A, Au TM, Brown FL, Bryant RA, Garcia-Moreno C, Musci RJ, Ventevogel P, White RG, van Ommeren M. Guided self-help to reduce psychological distress in South Sudanese female refugees in Uganda: a cluster randomised trial. Lancet Glob Health. 2020 Feb;8(2):e254-e263. doi: 10.1016/S2214-109X(19)30504-2. PMID 31981556
- [Background] Tortelli A, Perquier F, Melchior M, Lair F, Encatassamy F, Masson C, K'ourio H, Gourevitch R, Mercuel A. Mental Health and Service Use of Migrants in Contact with the Public Psychiatry System in Paris. Int J Environ Res Public Health. 2020 Dec 15;17(24):9397. doi: 10.3390/ijerph17249397. PMID 33333905
- [Background] Turrini G, Purgato M, Acarturk C, Anttila M, Au T, Ballette F, Bird M, Carswell K, Churchill R, Cuijpers P, Hall J, Hansen LJ, Kosters M, Lantta T, Nose M, Ostuzzi G, Sijbrandij M, Tedeschi F, Valimaki M, Wancata J, White R, van Ommeren M, Barbui C. Efficacy and acceptability of psychosocial interventions in asylum seekers and refugees: systematic review and meta-analysis. Epidemiol Psychiatr Sci. 2019 Aug;28(4):376-388. doi: 10.1017/S2045796019000027. Epub 2019 Feb 11. PMID 30739625
- [Background] United Nations. Policy Brief: Covid-19 and the Need for Action on Mental Health [Internet]. Geneva; 2020. Available from: https://unsdg.un.org/sites/default/files/2020-05/UN-Policy-Brief-COVID-19-and-mental-health.pdf
- [Background] University of Kent. The Unit Costs of Health and Social Care [Internet]. 2003. Available from: http://kar.kent.ac.uk/26657/
- [Background] Usher K, Bhullar N, Durkin J, Gyamfi N, Jackson D. Family violence and COVID-19: Increased vulnerability and reduced options for support. Int J Ment Health Nurs. 2020 Aug;29(4):549-552. doi: 10.1111/inm.12735. Epub 2020 May 7. No abstract available. PMID 32314526
- [Background] van Spijker BA, Batterham PJ, Calear AL, Farrer L, Christensen H, Reynolds J, Kerkhof AJ. The suicidal ideation attributes scale (SIDAS): Community-based validation study of a new scale for the measurement of suicidal ideation. Suicide Life Threat Behav. 2014 Aug;44(4):408-19. doi: 10.1111/sltb.12084. Epub 2014 Feb 24. PMID 24612048
- [Background] van Straten A, Hill J, Richards DA, Cuijpers P. Stepped care treatment delivery for depression: a systematic review and meta-analysis. Psychol Med. 2015 Jan;45(2):231-46. doi: 10.1017/S0033291714000701. Epub 2014 Mar 26. PMID 25065653
- [Background] van 't Hof E, Heim E, Abi Ramia J, Burchert S, Cornelisz I, Cuijpers P, El Chammay R, Harper Shehadeh M, Noun P, Smit F, van Klaveren C, van Ommeren M, Zoghbi E, Carswell K. Evaluating the Effectiveness of an E-Mental Health Intervention for People Living in Lebanon: Protocol for Two Randomized Controlled Trials. JMIR Res Protoc. 2021 Jan 28;10(1):e21585. doi: 10.2196/21585. PMID 33507158
- [Background] Veer IM, Riepenhausen A, Zerban M, Wackerhagen C, Puhlmann LMC, Engen H, Kober G, Bogemann SA, Weermeijer J, Uscilko A, Mor N, Marciniak MA, Askelund AD, Al-Kamel A, Ayash S, Barsuola G, Bartkute-Norkuniene V, Battaglia S, Bobko Y, Bolte S, Cardone P, Chvojkova E, Damnjanovic K, De Calheiros Velozo J, de Thurah L, Deza-Araujo YI, Dimitrov A, Farkas K, Feller C, Gazea M, Gilan D, Gnjidic V, Hajduk M, Hiekkaranta AP, Hofgaard LS, Ilen L, Kasanova Z, Khanpour M, Lau BHP, Lenferink DB, Lindhardt TB, Magas DA, Mituniewicz J, Moreno-Lopez L, Muzychka S, Ntafouli M, O'Leary A, Paparella I, Poldver N, Rintala A, Robak N, Rosicka AM, Roysamb E, Sadeghi S, Schneider M, Siugzdaite R, Stantic M, Teixeira A, Todorovic A, Wan WWN, van Dick R, Lieb K, Kleim B, Hermans EJ, Kobylinska D, Hendler T, Binder H, Myin-Germeys I, van Leeuwen JMC, Tuscher O, Yuen KSL, Walter H, Kalisch R. Psycho-social factors associated with mental resilience in the Corona lockdown. Transl Psychiatry. 2021 Jan 21;11(1):67. doi: 10.1038/s41398-020-01150-4. PMID 33479211
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] World Health Organisation. Measuring Health and Disability. Manual for WHO Disability Assessment Schedule (WHODAS 2.0) [Internet]. Geneva; 2010. Available from: https://apps.who.int/iris/handle/10665/43974
- [Background] World Health Organization. in the COVID-19 response in the WHO European Region Vulnerable populations during COVID-19 response [Internet]. Geneva; 2020. Available from: https://www.euro.who.int/__data/assets/pdf_file/0003/446340/Factsheet-May-2020-Vulnerable-populations-during-COVID-19-response-eng.pdf
- [Derived] Melchior M, Figueiredo N, Roversi A, Dubanchet A, Bui E, Vadell-Martinez J, Barbui C, Purgato M, Ayuso-Mateos JL, Mediavilla R, McDaid D, Park AL, Petri-Romao P, Kalisch R, Nicaise P, Lorant V, Sijbrandij M, Witteveen AB, Bryant R, Felez M, Underhill J, Pollice G, Tortelli A. Addressing mental health problems among persons without stable housing in the context of the COVID-19 pandemic: study protocol for a randomised trial. RESPOND - France. BMC Public Health. 2023 Nov 17;23(1):2275. doi: 10.1186/s12889-023-17238-7. PMID 37978577